CLINICAL TRIAL: NCT03162900
Title: A PHASE 1, SINGLE CENTER, RANDOMIZED, 4-WAY CROSSOVER, DOUBLE BLINDED, PLACEBO AND MOXIFLOXACIN CONTROLLED STUDY TO EVALUATE THE EFFECT OF GLASDEGIB ON THE CARDIAC REPOLARIZATION IN HEALTHY SUBJECTS
Brief Title: A Phase 1 Study To Evaluate The Effect Of Glasdegib On The Cardiac Repolarization In Healthy Subjects
Acronym: B1371023
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B1371023; 2017-001295-38 (EudraCT Number)
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers
Keywords: Glasdegib; PF-04449913; Pharmacokinetics; QTc; TQT
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glasdegib QT Therapeutic Exposure (Experimental): Randomized sequence of Glasdegib clinical exposure, Placebo and moxifloxacin active control administration. This treatment will be in four separate sequences with four periods per sequence. Each period will be separated by a washout of atleast 6 days.
  Interventions: Drug: Glasdegib Therapeutic Exposure; Drug: Positive Control (Moxifloxacin); Other: Placebo Control
- Glasdegib QT Supra-therapeutic Exposure (Experimental): Randomized sequence of glasdegib supra-therapeutic exposure, Placebo and moxifloxacin active control administration. This treatment will be in four separate sequences with four periods per sequence. Each period will be separated by a washout of atleast 6 days.
  Interventions: Drug: Glasdegib Supra-therapeutic Exposure

INTERVENTIONS:
Drug: Glasdegib Therapeutic Exposure — Subjects Receive a single 150 mg dose of Glasdegib followed by ECG and PK assessments.
  Arms: Glasdegib QT Therapeutic Exposure
Drug: Glasdegib Supra-therapeutic Exposure — Subjects receive a single 300 mg dose of glasdegib followed by ECG and PK assessments.
  Arms: Glasdegib QT Supra-therapeutic Exposure
Drug: Positive Control (Moxifloxacin) — Subjects will receive a single 400 mg dose of moxifloxacin followed by ECG and PK assessments.
  Arms: Glasdegib QT Therapeutic Exposure
Other: Placebo Control — Subjects will receive placebo dose followed by ECG and PK assessments.
  Arms: Glasdegib QT Therapeutic Exposure

SUMMARY:
This is a Thorough QT study intended to estimate the effect of glasdegib at therapeutic exposure and at supra-therapeutic exposure on cardiac repolarization in healthy subjects. This is a randomized, double blind, positive and placebo controlled study with a 6 day washout between successive periods.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy male and/or female subjects of non child bearing potential who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG or clinical laboratory tests.

Female subjects of nonchildbearing potential must meet at least 1 of the following criteria:

1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; with a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
3. Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy, bilateral oophorectomy and/or ovarian failure) are considered to be of childbearing potential.

   2. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

   3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

   4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

   Exclusion Criteria:
   * Screening supine 12 lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.

   Subjects with family history of myocardial infarction, congenital long QT syndrome, torsades de pointes or clinically significant ventricular arrhythmias. Subjects should be within normal range of potassium, magnesium and corrected calcium calculation at screening.

   Pregnant female subjects; breastfeeding female subjects; female subjects of childbearing potential; male subjects with partners currently pregnant; male subjects who are unwilling or unable to use atleast one highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 90 days after the last dose of investigational product and, refrain from sperm donation for the duration of the Study and for at least 90 days after the last dose of investigational product.

   History of known QTc prolongation or ECG abnormalities.

   Self-reported history of risk factors for QT prolongation or torsades de pointes (eg, organic heart disease, congestive heart failure, hypokalemia, hypomagnesemia,congenital long QT syndrome, myocardial ischemia or infarction, congenital deafness, and family history of sudden death, or a family history of congenital QT syndrome).

   Self-reported history of sick sinus syndrome, first, second, or third degree atrioventricular (AV) block, myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QT interval or conduction abnormalities, or any other clinically significant cardiovascular disease history.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2017-09-23 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
QTcF interval | 120 hours per period
  Post-dose placebo corrected QTcF intervals from ECG traces following glasdegib dosing.

SECONDARY OUTCOMES:
QTcF interval (Moxifloxacin) | 120 hours
  Post-dose placebo corrected QTcF intervals from ECG traces following moxifloxacin dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Masters JC, Shaik N, Mendes da Costa L, Hee B, LaBadie RR. Clinical and Model-Based Evaluation of the Effect of Glasdegib on Cardiac Repolarization From a Randomized Thorough QT Study. Clin Pharmacol Drug Dev. 2021 Mar;10(3):272-282. doi: 10.1002/cpdd.862. Epub 2020 Aug 12. PMID 32790066
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1371023